CLINICAL TRIAL: NCT01345097
Title: A Short Metaphyseal Fitting Total Hip Arthroplasty in Young and Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Young Hoo Kim, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: THRProxima
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Osteonecrosis; Osteoarthritis
Keywords: short, metaphyseal-fitting femoral stem; cementless anatomical femoral stem; young patient; elderly patient
MeSH Terms: conditions — Osteonecrosis; Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Younger Group (Experimental)
  Interventions: Device: Total Hip Arthroplasty
- Elderly Group (Experimental)
  Interventions: Device: Total Hip Arthroplasty

INTERVENTIONS:
Device: Total Hip Arthroplasty — Total Hip Arthroplasty
  Other Names: Proxima

SUMMARY:
The investigators determined whether

1. new short, metaphyseal-fitting cementless anatomical femoral stem provides major functional improvements
2. radiographically secure implant fixation is achieved with this new stem
3. the bone content is preserved at the baseline level or above at the final follow-up
4. these procedures are associated with early failure and complications.

DETAILED DESCRIPTION:
To attempt reduction of stress shielding and thigh pain as well as to improve survivorship, a new short, metaphyseal-fitting cementless anatomical femoral stem was developed. The question arises as to whether it is possible to obtain rigid fixation of the stem without diaphyseal fixation in the young as well as in the elderly patients. The purpose of this study was to determine the clinical and radiographic results of the new short, metaphyseal-fitting cementless anatomical femoral stem in the young as well as in the elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of hip joint requiring total hip arthroplasty

Exclusion Criteria:

* Neurologic disorders affecting motor function of lower extremity foot and ankle disorders limiting ambulation of the patient
* Patients with bone metabolic disorders other than osteoporosis which prevents normal bone metabolism
* Multi-systemic inflammatory arthritis which debilitates patients other than hip joint.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-05; Primary Completion 2006-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Harris hip score | At least 5 years after surgery
  This is a verified scoring tool for measuring hip function.

SECONDARY OUTCOMES:
Improvement in the Range of Motion | At least 5 years after surgery
  The change in the hip range motion compared to the initial and the last measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoo Kim, MD, Study Director — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha Womans University Mokdong Hosptial, Seoul, South Korea